CLINICAL TRIAL: NCT05086380
Title: Modulation of the Sense of Agency Across Different Neurological Disorders Using Non-invasive Brain Stimulation and Mindfulness-based Stress Reduction Therapy
Brief Title: Modulation of Sense of Agency With Non-invasive Brain Stimulation and Mindfulness-based Stress Reduction Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Fribourg (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-02283
Record Dates: First submitted 2021-09-10; First posted 2021-10-20 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Functional Neurological Symptom Disorder; Neurological Diseases or Conditions
MeSH Terms: conditions — Conversion Disorder | interventions — Mindfulness-Based Stress Reduction; Neurofeedback

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FND Patients Experimental (Experimental): Group of patients with functional neurological disorders
  Interventions: Behavioral: Mindfulness-based stress reduction therapy; Device: Inhibitory TMS; Device: TMS sham; Device: Excitatory TMS; Device: Virtual Reality; Behavioral: Neurofeedback
- Organic controls (Active Comparator): Group of patients with organic neurological disorders
  Interventions: Device: Inhibitory TMS; Device: TMS sham; Device: Excitatory TMS
- Healthy controls (Active Comparator): Group of healthy controls
  Interventions: Device: Inhibitory TMS; Device: TMS sham; Device: Excitatory TMS; Device: Virtual Reality
- FND Patients Comparator (Active Comparator): Group of patients with functional neurological disorders
  Interventions: Device: Inhibitory TMS; Behavioral: Psychoeducation; Device: TMS sham; Device: Excitatory TMS; Behavioral: Neurofeedback

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction therapy — MBSR Therapy is a structured 8-week program that employs mindfulness meditation to alleviate suffering associated with physical, psychosomatic and psychiatric disorders. The program is based upon a systematic procedure to develop enhanced awareness of moment-to-moment experience of perceptible mental processes.
  Arms: FND Patients Experimental
Device: Inhibitory TMS — The device will be used to neuromodulate the right TPJ of participants' brain using cTBS stimulation protocol for transcranial magnetic stimulation
Behavioral: Psychoeducation — Participants will learn about the symptoms and how to cope with the symptoms
  Arms: FND Patients Comparator
Device: TMS sham — The device will be used to neuromodulate the right TPJ of participants' brain using transcranial magnetic stimulation over the vertex
Device: Excitatory TMS — The device will be used to neuromodulate the right TPJ of participants' brain using iTBS stimulation protocol for transcranial magnetic stimulation
Device: Virtual Reality — The device will be used to manipulate the perception of symptoms of patients while they are playing a game in virtual/augmented reality.
  Arms: FND Patients Experimental; Healthy controls
Behavioral: Neurofeedback — Neurofeedback training will be applied in patients while laying in an MRI scanner. Patients will play a game, which targets the sense of agency, and will receive a real-time feedback about their performance and brain activity. They will learn to self-regulate their performance on the game in order to increase brain activity relevant for the sense of agency.
  Arms: FND Patients Comparator; FND Patients Experimental

SUMMARY:
A conversion disorder is a dysfunction of the nervous system in which no structural damage can be demonstrated. However, it must be distinguished from other psychiatric disorders such as psychosis or depression. There are a variety of signs of the disease, such as muscle paralysis, uncontrolled tremors or cramps. In rarer cases, blindness, deafness or numbness may occur. Diagnosing this complex disorder has always been a challenge for neurologists and psychiatrists.

This study investigates the effects of transcranial magnetic stimulation (TMS) on the general well-being and symptoms of conversion disorder and other neurological disorders and in comparison to healthy subjects. The TMS method allows to target specific areas of the brain by means of magnetic fields. This technique is not painful and does not have long-lasting effects.

In addition, the study investigates the effects of mindfulness-based stress reduction on the general well-being and symptoms of conversion disorder and other neurological disorders and compared to healthy subjects. This technique is not painful and has no long-lasting effects.

Furthermore, the study examines movement patterns and symptoms of patients compared to healthy controls while they are in a virtual reality.

Finally, the study examines patients' brain activity while playing a game targeting the sense of agency in real time, which is recorded with an MRI scanner.

The study includes a maximum of twelve sessions in total (ten sessions of approximately 1.5-2 hours each and two sessions each overnight). The planned study methods include TMS, (real-time and normal) magnetic resonance tomography of the brain (MRI "tube"), virtual- and augmented reality (AR/VR), questionnaires, blood, saliva, and motion sensors (e.g., fitness bracelet), and participation in the 8-week mindfulness program.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* A diagnosis of a functional disorder (such as FND, GTS, PPD, anxiety or depression or others) according to DSM-5 diagnostic and ICD-11 criteria, or
* A diagnosis of an organic neurological disorder such as stroke, multiple sclerosis (MS), neuromuscular, or movement disorder
* Aged > 16 years old
* Willing to participate in the study (by signing the ICF)
* Capable of judgement

healthy controls:

* Aged > 16 years old
* Willing to participate in the study (by signing the ICF)
* Capable of judgement

Exclusion Criteria:

* Presence of comorbid psychiatric disorders such as psychosis, current major and severe depression episode, autistic spectrum disorder
* Past surgery in the brain
* History of alcohol or drug abuse
* Botulinum toxin injection in last 3 month
* Inability to follow the procedure of the study, e.g., due to language problems
* For organic disorders only: Active severe aphasia, dementia, neglect and acute confusional state, severe pain
* For female participants: breastfeeding, pregnancy or intention to become pregnant (assessed with standard urine test prior to the enrolment in the experiment and before each visit)
* For MRI and TMS part only: Past surgery in the brain
* For MRI and TMS part only: Implanted medical devices not-compatible with MRI or TMS (e.g., cochlear implants, infusion pumps, neurostimulators, cardiac pacemakers)
* For TMS part only: History of actual or suspected epilepsy
* For TMS part only: Suspected or diagnosed labile or hypertensive blood pressure
* For Virtual Reality only: No cybersickness

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Change in objective Performance Agency Task (TMS) | Visit 1 (at baseline), visit 2 (one week after baseline), visit 3 (two weeks after baseline), visit 7 to 11 (12 - 16 weeks)
  The changes in objective performance on the behavioural tasks targeting the sense of agency using the score of an agency task played in the Magnetic Resonance Imaging (MRI) scanner, on a computer or in Virtual Reality before and after brain stimulation (transcranial magnetic stimulation, TMS). The performance is measured by counting the number of targets hit minus the number of obstacles hit during the computer game [-].
Change in subjective Performance Agency Task (TMS) | Visit 1 (at baseline), visit 2 (one week after baseline), visit 3 (two weeks after baseline), visit 7 to 11 (12 - 16 weeks)
  The changes in objective and subjective performance on the behavioural tasks targeting the sense of agency using questionnaires before and after brain stimulation. Participants rate their performance on a visual analog scale (VAS) from 0 to 10 [-].
Change in objective Performance Agency Task (MBSR) | Visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4), visit 7 to 11 (12 - 16 weeks)
  The objective performance on the behavioural tasks targeting the sense of agency using the score of an agency task played in the MRI scanner, on a computer or in Virtual Reality before and after a therapeutic intervention (mindfulness-based stress reduction, MBSR).The performance is measured by counting the number of targets hit minus the number of obstacles hit during the computer game [-].
Change in subjective Performance Agency Task (MBSR) | Visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4), visit 7 to 11 (12 - 16 weeks)
  The subjective performance on the behavioural tasks targeting the sense of agency using questionnaires before and after a therapeutic intervention (MBSR). Participants rate their performance on a visual analog scale (VAS) from 0 to 10 [-].

SECONDARY OUTCOMES:
task-based fMRI measures TMS | Visit 1 (at baseline), visit 2 (one week after baseline), visit 3 (two weeks after baseline)
  The functional magnetic resonance imaging (fMRI) measures of blood oxygenation signal (BOLD) in the whole brain during the behavioural task before and after excitatory, inhibitory or sham rTMS, in patients affected by a functional neuropsychiatric disorder (e.g., FND, Gilles de la Tourette Syndrome (GTS), Psychosomatic Pain Disorder (PPD)), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke) and healthy subjects. BOLD is measured in change in intensity between conditions with conditions being before and after rTMS [-].
resting-state fMRI measures TMS | Visit 1 (at baseline), visit 2 (one week after baseline), visit 3 (two weeks after baseline)
  The fMRI measures of blood oxygenation in the whole brain at rest, before and after excitatory, inhibitory or sham rTMS, in patients affected by a functional neuropsychiatric disorder (e.g., FND, GTS, PPD), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke) and healthy subjects. BOLD is measured in change in functional connectivity between conditions with conditions being before and after rTMS. Functional connectivity is calculated using Pearson's correlation coefficient between pairs of brain regions [-].
DTI measures TMS | Visit 1 (at baseline), visit 2 (one week after baseline), visit 3 (two weeks after baseline)
  The fMRI measures of blood oxygenation in the whole brain using diffusion tensor imaging (DTI), before and after excitatory, inhibitory or sham rTMS, in patients affected by a functional neuropsychiatric disorder (e.g., FND, GTS, PPD), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke) and healthy subjects. DTI measures the direction and strengths of white matter fibre tracts by measuring the diffusion of water molecules. The measured quantity is the diffusivity or diffusion coefficient, a proportionality constant that relates diffusive flux to a concentration gradient [mm2/s].
task-based fMRI measures MBSR | Visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4)
  The fMRI measures of blood oxygenation in the whole brain during the behavioural task, before and after MBSR or psychoeducation, in patients affected by a functional neuropsychiatric disorder (e.g., FND, GTS, PPD), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke). BOLD is measured in change in intensity between conditions with conditions being before and after rTMS [-].
resting-state fMRI measures MBSR | Visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4)
  The fMRI measures of blood oxygenation in the whole brain at rest before and after MBSR or psychoeducation, in patients affected by a functional neuropsychiatric disorder (e.g., FND, GTS, PPD), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke). BOLD is measured in change in functional connectivity between conditions with conditions being before and after rTMS. Functional connectivity is calculated using Pearson's correlation coefficient between pairs of brain regions [-].
DTI measures MBSR | Visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4)
  The fMRI measures of blood oxygenation in the whole brain during DTI, before and after MBSR or psychoeducation, in patients affected by a functional neuropsychiatric disorder (e.g., FND, GTS, PPD), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke). DTI measures the direction and strengths of white matter fibre tracts by measuring the diffusion of water molecules. The measured quantity is the diffusivity or diffusion coefficient, a proportionality constant that relates diffusive flux to a concentration gradient [mm2/s].
Subjective Agency TMS | Visit 1 (at baseline), visit 2 (one week after baseline), visit 3 (two weeks after baseline)
  Subjective assessment of own agency during a behavioural task, before and after excitatory, inhibitory or sham rTMS, in patients affected by a functional neuropsychiatric disorder (e.g., FND, Gilles de la Tourette Syndrome (GTS), Psychosomatic Pain Disorder (PPD)), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke) and healthy subjects. Participants rate their performance on a visual analog scale (VAS) from 0 to 10 [-].
Subjective Agency MBSR | Visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4)
  Subjective assessment of own agency during a behavioural task, before and after MBSR or psychoeducation, in patients affected by a functional neuropsychiatric disorder (e.g., FND, GTS, PPD), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke). Participants rate their performance on a visual analog scale (VAS) from 0 to 10 [-].
Neurological Examination TMS | Visit 1 (at baseline), visit 2 (one week after baseline), visit 3 (two weeks after baseline)
  The performance on an objective neurological examination, before and after excitatory, inhibitory or sham rTMS, in patients affected by a functional neuropsychiatric disorder (e.g., FND, Gilles de la Tourette Syndrome (GTS), Psychosomatic Pain Disorder (PPD)), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke). Patients will be examined according to standardized medical examination tests (e.g., positive signs & A Simplified Version of the Psychogenic Movement Disorders Scale (S-FMDRS) for FND).
Neurological Examination MBSR | Visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4)
  The performance on an objective neurological examination, before and after MBSR or psychoeducation in patients affected by a functional neuropsychiatric disorder (e.g., FND, GTS, PPD), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke). Patients will be examined according to standardized medical examination tests (e.g., positive signs & A Simplified Version of the Psychogenic Movement Disorders Scale (S-FMDRS) for FND).
Objective stress parameters pre/post | Visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4)
  The stress parameters assessed using salivary cortisol before and after MBSR Therapy compared to psychoeducation, in patients affected by a functional neuropsychiatric disorder, an organic condition or in healthy subjects. Cortisol levels are measured using Enzyme-linked Immunosorbent Assay (ELISA) [ng/ul].
Subjective stress parameters pre/post | Visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4)
  Subjective stress before and after MBSR Therapy compared to psychoeducation, in patients affected by a functional neuropsychiatric disorder, an organic condition or in healthy subjects. Subjective stress is measured using a VAS from 0-100.
Sleep | Visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4)
  The outcomes of ambient sensors (i.e., actigraphs) monitor non-invasively everyday life activity (ELA), including sleep, in patients affected by a functional neuropsychiatric disorder, an organic condition or in healthy subjects. Actigraphs measure light input and motion. A variety of outcome measures can be calculated such as Time in Bed, Time asleep,
Neurofeedback | Visit 7 to 11 (12 - 16 weeks)
  The real-time measures of blood oxygenation in the target areas (e.g., TPJ) in patients affected by a functional neuropsychiatric disorder (e.g., FND, GTS, PPD), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke) and healthy subjects. Participants will receive direct feedback on their performance in the scanner.
Long-term effects on task-based fMRI measures MBSR | At follow-up (6 month after visit 5)
  To measure the long-term (six months) effect of MBSR Therapy, the fMRI measures of blood oxygenation signal (BOLD) is measured in the whole brain during the behavioural task, in patients affected by a functional neuropsychiatric disorder (e.g., FND, Gilles de la Tourette Syndrome (GTS), Psychosomatic Pain Disorder (PPD)), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke) and healthy subjects. BOLD is measured in change in intensity between conditions with conditions being at follow-up compared to Visit 5 (after MBSR therapy)[-].
Long-term effects on resting-state fMRI measures MBSR | At follow-up (6 month after visit 5)
  To measure the long-term (six months) effect of MBSR Therapy, the fMRI measures of blood oxygenation signal (BOLD) is measured in the whole brain at rest, in patients affected by a functional neuropsychiatric disorder (e.g., FND, GTS, PPD), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke) and healthy subjects. BOLD is measured in change in functional connectivity between conditions with conditions being at follow-up compared to Visit 5 (after MBSR therapy). Functional connectivity is calculated using Pearson's correlation coefficient between pairs of brain regions [-]. .
Long-term effects on DTI measures MBSR | At follow-up (6 month after visit 5)
  To measure the long-term (six months) effect of MBSR Therapy, the fMRI measures of blood oxygenation signal (BOLD) is measured in the whole brain during DTI, in patients affected by a functional neuropsychiatric disorder (e.g., FND, GTS, PPD), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke) and healthy subjects. DTI measures the direction and strengths of white matter fibre tracts by measuring the diffusion of water molecules. The measured quantity is the diffusivity or diffusion coefficient, a proportionality constant that relates diffusive flux to a concentration gradient [mm2/s].
Long-term effects on subjective agency MBSR | At follow-up (6 month after visit 5)
  To measure the long-term (six months) effect of MBSR therapy, the subjective performance on the behavioural tasks targeting the sense of agency is used. Participants rate their agency on a visual analog scale (VAS) from 0 to 10 [-]. Subjective agency at follow-up will be compared to subjective agency at Visit 5 (after MBSR).
Long-term effects on neurological examination MBSR | At follow-up (6 month after visit 5)
  To measure the long-term (six months) effect of MBSR therapy, the performance on an objective neurological examination will be assessed, in patients affected by a functional neuropsychiatric disorder (e.g., FND, GTS, PPD), in comparison to patients affected by an organic condition (e.g., Dystonia, Stroke). Patients will be examined according to standardized medical examination tests (e.g., positive signs & A Simplified Version of the Psychogenic Movement Disorders Scale (S-FMDRS) for FND). Outcome of neurological assessment at follow-up will be compared to outcome of neurological assessment at Visit 5 (after MBSR).
Long-term effects on objective performance | At follow-up (6 month after visit 5)
  To measure the long-term (six months) effect of MBSR therapy, the objective performance on the behavioural tasks targeting the sense of agency is used. The performance is measured by counting the number of targets hit minus the number of obstacles hit during the computer game [-]. Objective performance at follow-up will be compared to objective performance at Visit 5 (after MBSR).
Long-term effects on subjective performance | At follow-up (6 month after visit 5)
  To measure the long-term (six months) effect of MBSR therapy, the subjective performance on the behavioural tasks targeting the sense of agency is used. Participants rate their performance on a visual analog scale (VAS) from 0 to 10 [-]. Objective performance at follow-up will be compared to objective performance at Visit 5 (after MBSR).
Neurophysiological measures: MEP | Visit 1 (at baseline), visit 2 (one week after baseline), visit 3 (two weeks after baseline), visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4) and follow up (6 month after visit 5)
  Motor evoked potential (MEP) is measured by eliciting an action potential using non-invasive brain stimulation (TMS) over the motor cortex through the scalp [% TMS - max. intensity output]. Neurophysiological measures will be used to characterise movement disorders. We will compare MEPs in patients with a functional, or organic condition, to healthy subjects.
Neurophysiological measures: MT | Visit 1 (at baseline), visit 2 (one week after baseline), visit 3 (two weeks after baseline), visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4) and follow up (6 month after visit 5)
  Motor threshold (MT) measures the intensity of a pulse which elicits a predefined MEP. Neurophysiological measures will be used to characterise movement disorders. We will compare MTs in patients with a functional, or organic condition, to healthy subjects.
Neurophysiological measures: SICI | Visit 1 (at baseline), visit 2 (one week after baseline), visit 3 (two weeks after baseline), visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4) and follow up (6 month after visit 5)
  Short IntraCortical Inhibition (SICI) measures the reduction of the MEP occurring after weak (subthreshold) conditioning pulse followed by a supra-threshold test pulse at short interstimulus intervals (approximately 2 msec). Neurophysiological measures will be used to characterise movement disorders. We will compare SICIs in patients with a functional, or organic condition, to healthy subjects.
Neurophysiological measures: LICI | Visit 1 (at baseline), visit 2 (one week after baseline), visit 3 (two weeks after baseline), visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4) and follow up (6 month after visit 5)
  Long IntraCortical Inhibition (LICI) measures the reduction of MEP, as described in Outcome 28, at long interstimulus intervals (between 50 and 200 msec), using supra-threshold paired stimulation. Neurophysiological measures will be used to characterise movement disorders. We will compare LICIs in patients with a functional, or organic condition, to healthy subjects.
Neurophysiological measures CSP | Visit 1 (at baseline), visit 2 (one week after baseline), visit 3 (two weeks after baseline), visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4) and follow up (6 month after visit 5)
  Cortical Silent Period (CSP) measures the period of electromyography (EMG) silence before activity resumes baseline, following the MEP elicited by a pulse to the motor cortex during tonic contraction of a target muscle. Neurophysiological measures will be used to characterise movement disorders. We will compare CSPs in patients with a functional, or organic condition, to healthy subjects.
Neurophysiological measures: PAS | Visit 1 (at baseline), visit 2 (one week after baseline), visit 3 (two weeks after baseline), visit 4 (at least 1 week after visit 3), visit 5 (8 weeks after visit 4) and follow up (6 month after visit 5)
  Paired Associative Stimulation (PAS) measures the increase in the MEP amplitude following lowfrequency stimulation over the median nerve of the hand, paired with TMS over the motor cortex. This is an index for plasticity. Neurophysiological measures will be used to characterise movement disorders. We will compare CSPs in patients with a functional, or organic condition, to healthy subjects.
Epigenetic profile | 1st visit (baseline)
  Mean methylation rates of genes involved in the stress-pathway (i.e., Oxytocin, Serotonine, Dopamine, Glucocorticoid receptor) will be assessed in patients affected by a functional or organic disorder and healthy subjects using blood samples. Methylation profiles will be determined using the bisulfite - treatment method.
Long-term fluctuations of objective stress parameters | at follow-up (6 month after visit 5)
  To assess the long-term (six months) fluctuations of stress, salivary cortisol will be measured at follow-up in patients affected by a functional neuropsychiatric disorder, an organic condition or in healthy subjects. Cortisol levels are measured using Enzyme-linked Immunosorbent Assay (ELISA) [ng/ul].
Long-term fluctuations of subjective stress parameters | at follow-up (6 month after visit 5)
  To assess the long-term (six months) fluctuations of stress, subjective stress levels will be measured at follow-up in patients affected by a functional neuropsychiatric disorder, an organic condition or in healthy subjects. Subjective stress is measured using a VAS from 0-100.
Position of focus of attention | at visit 6 (at least one week after visit 5)
  To assess the position of focus of attention we will use eye tracking while participants play a game in virtual reality. We assess where participants focus their attention while moving their limbs
Kinematics of limb movements | at visit 6 (at least one week after visit 5)
  To assess the kinematics of movements of participants, we apply motion tracking systems with which we measure movement translation and rotation in space.
Stability | Visit 1 (at baseline), and follow up (8 month after visit 1)
  The objective and subjective sway in functional patients, organic control patients and healthy subjects will be assessed using posturography, which includes diverse balance exercises on a force plate (e.g. with eyes open / with eyes closed).
Cognition | Visit 1 (at baseline), and follow up (8 month after visit 1)
  Outcomes of neuropsychiatric test battery will be compared in functional patients, organic control patients and healthy subjects (e.g. attention, working memory), and further correlated with the fMRI BOLD signal in e.g., the multimodal vestibular network.
Pain processing | Visit 1 (at baseline), and follow up (8 month after visit 1)
  Pain processing and perception of pain will be studied in functional patients, organic patients and healthy subjects by using a standardized tool (i.e. Algopeg). Scores from Algopeg will be associated with neural correlates (e.g., resting state fMRI).

CONTACTS AND LOCATIONS:
Overall Officials: Selma Aybek, MD, Principal Investigator — University of Fribourg
Locations (1):
- University of Fribourg, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No